CLINICAL TRIAL: NCT01298024
Title: NEMEX-ATR: A Randomized Pilot Study on Early Neuromuscular Exercise in Non-surgically Treated Achilles Tendon Rupture
Brief Title: A Pilot Study on Exercise After Achilles Tendon Rupture
Acronym: NEMEX-ATR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/173
Record Dates: First submitted 2011-02-09; First posted 2011-02-17 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture; Non-surgical treatment; Exercise; Neuromuscular training
MeSH Terms: conditions — Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early neuromusclar exercise (Experimental)
  Interventions: Other: Early Neuromuscular Exercise
- Treatment as usual (late training) (Active Comparator)
  Interventions: Other: Early Neuromuscular Exercise

INTERVENTIONS:
Other: Early Neuromuscular Exercise — 30 patients are randomized to early neuromuscular exercise (n=15) or treatment as usual, i.e., late exercise (n=15). Both groups are given an orthosis and are instructed to wear this for eight weeks. The experimental group starts with a structured exercise program one week after the diagnosis. The patients attend one training session/week during eight weeks, guided by a physical therapist. The level of training is progressed during this time. The patients in the control group (treatment as usual) are given exercise instructions and information at one occasion; 2 weeks after diagnosis. Both groups are followed up, by a blinded assessor, with valid and reliable self-reported and physical function outcomes at 1, 4, 8 and 16 weeks after injury.
  Other Names: Treatment as usual (late exercise)

SUMMARY:
The purpose is to study the effect of early NEuroMuscular EXercise (NEMEX) versus conventional treatment (late exercise) in patients with acute non-operative achilles tendon rupture (ATR).

DETAILED DESCRIPTION:
There is currently no consensus on treatment for achilles tendon rupture with regard to surgical or non-surgical treatment. In addition, the optimal time to start exercise treatment after the injury, with or without surgery, is not well understood. Animal studies show positive effects of early mobilization in tendon healing. Neuromuscular exercise has shown better effects than strength exercise in people with knee injury or knee disease. There are few studies in humans focusing on exercise as treatment, without surgical intervention, after ATR.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 - 60 years.
2. The patient should before the achilles tendon rupture have been able to walk independently without aid, walk without limping, run/jog and be able to jump on one leg
3. The patient shall be able to read, understand and to assimilate the written information about the study.

Exclusion Criteria:

1. Previous achilles tendon rupture
2. Acute achilles tendon rupture, more than 5 days.
3. Medical restrictions regarding physical exercise, not related to the achilles tendon rupture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Heel-raise | Week 16
  Functional performance of calf muscles. The ability to perform a plantar flexion is assessed in a prone position at 1 and 4 weeks after the injury. At 8 and 16 weeks after the injury, the ability to perform a heel-raise standing on one leg is assessed.

SECONDARY OUTCOMES:
Single limb standing balance | At weeks 4, 8 and 16
  The patients stands on one leg with eyes open as long as possible, maximum time 60 seconds. Both legs are tested.
30-meters walk test | At weeks 8 and 16
  The patients walks a distance of 30 m at self-selected speed. Time and any limbing is recorded.
Single-limb mini squat | At week 16
  The patients performs single-limb mini squats. The position of the knee in relation to the foot is assessed. The test is performed on both legs.
VAS Pain | At weeks 1, 4, 8 and 16
  The patients reports pain on a 0-10 visual analog scale.
Range of Motion | At weeks 1, 4, 8 and 16
  The range of plantar and dorsal flexion motions in the talocrural joint are measured with a handheld goniometer.
The calf muscle circumference | At weeks 1, 4, 8 and 16
  Calf muscle circumference is recording using a measuring-tape.
Foot and Ankle Outcome Score (FAOS) | At weeks 1, 4, 8 and 16
  A disease specific questionnaire for patients with foot and ankle injury.
Short-Form 36 (SF-36) | At weeks 1, 4, 8 and 16
  A generic measure of health status.
Physical Activity Level Scale | At weeks 1, 4, 8 and 16
  A scale that measures the patient's level of daily physical activity.
Re-rupture | Weeks 1-16
  Joint specific adverse event; recorded by any patient seeking medical care related to the achilles tendon rupture during the study period.
Deep Venous thromboembolism | Weeks 1-16
  Joint specific adverse event; recorded by any patient seeking medical care related to the achilles tendon rupture during the study period.
Sick leave | Measured regularly from baseline until week 16
  The number of weeks the patient are not at work caused of the achilles tendon rupture is registered.
Modified Forward lunge from stairs | week 16
  The patient stands on the first step of a staircase and is encouraged to take step down with one leg, the other leg kept on the step. The examiner stands in front of the patient and observes position of joints in relation to each other.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PT, PhD, Study Director — Lund University; Sylvia Resch, MD, PhD, Study Director — Skane University Hospital
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden